CLINICAL TRIAL: NCT01269528
Title: Prospective Evaluation of the Efficacy of Palivizumab Administration in Children Born at 29-32 Weeks of Gestation
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: Evaluation of Palivizumab
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Bronchial Hyperreactivity; Infant, Premature
Keywords: Palivizumab; Airway Hyperreactivity; EBC; MCT
MeSH Terms: conditions — Bronchial Hyperreactivity; Premature Birth | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood for complete blood count , IGE and cytokines.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Born in 2007-2008: Methacholine Challenge Test (MCT). Monthly telephone contact. Visits to the study site. Fractional exhaled nitric oxide. Blood test.
  Interventions: Other: Methacholine Challenge Test (MCT); Other: Monthly telephone contact; Other: Visits to the study site; Other: Blood Test; Other: Fractional exhaled nitric oxide
- Born in 2009-2010: Methacholine Challenge Test (MCT). Monthly telephone contact. Visits to the study site. Fractional exhaled nitric oxide. Blood test.
  Interventions: Other: Methacholine Challenge Test (MCT); Other: Monthly telephone contact; Other: Visits to the study site; Other: Blood Test; Other: Fractional exhaled nitric oxide

INTERVENTIONS:
Other: Methacholine Challenge Test (MCT) — MCT challenge with determination of methacholine concentration that causes a 20% decrease from baseline FEV1 (forced expiratory volume in the 1st second of expiration) - PC20-FEV1 - is a well-documented method of assessing bronchial hyper-reactivity (BHR) in both adults and children. Our group has shown that the determination of PC20 by spirometry is feasible in preschool children. MCT is considered safe in this age group and our group has extensive experience with no adverse events. In the current study MCT will be performed (for the first time) in premature babies born at 30-32 weeks of gestation during 2008-2009 when they reach the age of 3-4 years (2011 and 2012, respectively). The results of MCT of the two groups will be compared.
Other: Monthly telephone contact — Monthly telephone contact with the parents/caregivers will be scheduled from enrollment until the final visit at age 3-4 years. Subject illnesses and other medical events occurring during the past month will be recorded at each monthly follow-up.
Other: Visits to the study site — Visits to the study site will be conducted at 6-month intervals in which physicians will record intercurrent doctor visits, emergency visits, and hospitalizations for respiratory symptoms.
Other: Blood Test — For assessing IgE levels, Eosinophils count and cytokines levels
Other: Fractional exhaled nitric oxide — Participant blow tidal volume for determination of exhaled NO in Exhaled breath.

SUMMARY:
Protocol Synopsis: There is a link between early RSV infection and chronic respiratory morbidity.

Hypothesis: Palivizumab administration may result in decreased AHR and lower respiratory morbidity.

Primary objective: to evaluate prospectively the effect of palivizumab on airway reactivity (AHR) in children born at 29-32 weeks.

Secondary objective: to assess prospectively the effect of palivizumab on respiratory morbidity airway inflammation and allergy in children born at 29-32 weeks.

Inclusion criteria: premature babies 29-32 weeks of gestation born during 2007 and 2010.

Exclusion criteria: Any mechanical ventilation or chronic diseases, e.g., bronchopulmonary dysplasia (BPD), cystic fibrosis (CF), congenital heart disease, congenital anomalies, known immunodeficiency, or receipt of other RSV investigative vaccines or therapies.

Primary end points: Airway reactivity as assessed by methacholine challenge test with determination of PC20.

Secondary end points: Respiratory morbidity as assessed by questionnaire and telephone interviews. Additionally, IGE, eosinophil count, and exhaled NO will be evaluated.

Sample size: 74 participants; Group I - 37 premature babies at 29-32 weeks of gestation born during 2007-2008 (before approval of Synagis for this group in Israel). Group II - 37 premature babies 29-32 weeks of gestation born during 2009-2010 (after approval of Synagis for this group in Israel).

Statistics: A sample size of 37 patients was calculated as necessary to detect a difference of 0.5 SD in AHR for a 2-sided tail, with a power of 80%. Demographics and baseline characteristics will be compared using 1-way analysis of variance for quantitative variables and Fisher's exact test for categorical variables.

DETAILED DESCRIPTION:
Protocol Synopsis: There is a link between early RSV infection and chronic respiratory morbidity.

Hypothesis: Palivizumab administration may result in decreased AHR and lower respiratory morbidity.

Primary objective: to evaluate prospectively the effect of palivizumab on airway reactivity (AHR) in children born at 29-32 weeks.

Secondary objective: to assess prospectively the effect of palivizumab on respiratory morbidity airway inflammation and allergy in children born at 29-32 weeks.

Inclusion criteria: premature babies 29-32 weeks of gestation born during 2007 and 2010.

Exclusion criteria: Any mechanical ventilation or chronic diseases, e.g., bronchopulmonary dysplasia (BPD), cystic fibrosis (CF), congenital heart disease, congenital anomalies, known immunodeficiency, or receipt of other RSV investigative vaccines or therapies.

Primary end points: Airway reactivity as assessed by methacholine challenge test with determination of PC20.

Secondary end points: Respiratory morbidity as assessed by questionnaire and telephone interviews. Additionally, IGE, eosinophil count, and exhaled NO will be evaluated.

Sample size: 74 participants; Group I - 37 premature babies at 29-32 weeks of gestation born during 2007-2008 (before approval of Synagis for this group in Israel). Group II - 37 premature babies 29-32 weeks of gestation born during 2009-2010 (after approval of Synagis for this group in Israel).

Statistics: A sample size of 37 patients was calculated as necessary to detect a difference of 0.5 SD in AHR for a 2-sided tail, with a power of 80%. Demographics and baseline characteristics will be compared using 1-way analysis of variance for quantitative variables and Fisher's exact test for categorical variables..

ELIGIBILITY:
Inclusion Criteria:

* Premature babies 29-32 weeks of gestation born during 2007 and 2010

Exclusion Criteria:

* Any mechanical ventilation
* Chronic diseases, e.g., bronchopulmonary dysplasia (BPD), cystic fibrosis (CF), congenital heart disease, congenital anomalies
* Known immunodeficiency
* Receipt of other RSV investigative vaccines or therapies

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature babies 29-32 weeks of gestation born during 2007 and 2010
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Airway reactivity | Between the 3 to 4 years-of-age
  As assessed by methacholine challenge test with determination of PC20 and inflammatory mediators in exhaled breath condensate.

SECONDARY OUTCOMES:
Respiratory morbidity | every month
  Monthly telephone contact with the parents/caregivers will be scheduled from enrollement until the final visit at age 3-4 years. Visits to the study site will be conducted at 6-month intervals. Subject illnesses and other medical events occurring during the past month will be recorded at each monthly follow-up. At 6-month intervals, physicians will record intercurrent doctor visits, emergency visits, and hospitalizations for respiratory symptoms.
IgE | Between the 3 to 4 years-of-age
  in pereferal Blood count
Eosinophil count | Between the 3 to 4 years-of-age
  in pereferal Blood count
skin tests for inhaled allergens | Between the 3 to 4 years-of-age

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel